CLINICAL TRIAL: NCT01893008
Title: Preoperative Inspiratory Muscle Training to Prevent Postoperative Pneumonia in Patients Undergoing Esophageal Resection
Brief Title: Preoperative Inspiratory Muscle Training in Esophageal Resection
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Frank JG Backx, MD PhD, Professor in Clinical Sports Medicine, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL43194.041.13
Record Dates: First submitted 2013-06-17; First posted 2013-07-08 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Resection Candidates
Keywords: Esophageal cancer; Surgery
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care + Inspiratory Muscle Training (IMT) (Experimental)
  Interventions: Other: Inspiratory Muscle Training (IMT)
- Usual care (no IMT) (No Intervention)

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) — The IMT protocol is tailored individually. Inspiratory load is set at 60% of the measured maximal inspiratory pressure (Pimax). The load is incrementally increased based on the rate of perceived exertion (RPE) scored on a scale from 0 to 10 which is scored by the patient after each training session. When patients score an RPE below 7, patients increase the inspiratory load of the threshold device with 5% to guarantee overload during each training session. Patients have to complete 30 dynamic inspiratory efforts twice daily.
  Patients will be instructed to train at home 7 days a week until surgery with a minimum of 2 weeks.
  Training will be started after the chemoradiation period (if applicable).
  Arms: Usual care + Inspiratory Muscle Training (IMT)

SUMMARY:
The PREPARE study is the first multicenter randomized controlled trial to evaluate the hypothesis that preoperative inspiratory muscle training leads to decreased pulmonary complications in patients undergoing esophageal resection.

DETAILED DESCRIPTION:
Rationale: Esophageal resection is associated with high incidences of postoperative pulmonary pneumonia. Numbers of 30% are reported in literature. Postoperative complications can result in prolonged hospital stay and increased health care costs. In cardiac surgery patients a reduction of postoperative pneumonia of 50% is reported as a result of a preoperative inspiratory muscle training program. While in some surgical centers IMT is already used in the preoperative phase in patients undergoing esophageal resection, the effect of this promising intervention has not yet been investigated in a randomised and controlled study design in large surgical populations other than cardiac surgery.

Primary objective: Investigate the effect of a preoperative inspiratory muscle training program on the incidence of postoperative pneumonia in patients undergoing esophageal resection.

Study design: Prospective multicenter randomised controlled clinical trial.

Main study parameters/endpoints: A significant reduction in incidence of postoperative pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* (Cognitively) capable to understand and perform a preoperative IMT program
* Surgery is scheduled at least 2 weeks after signing informed consent, since the patients need to be able to follow the intervention program for at least 2 weeks
* Willing to sign the informed consent form

Exclusion Criteria:

* Unable to communicate in Dutch language
* Age < 18 years
* Participating in a conflicting trial concerning esophageal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pneumonia incidence | Date of first pneumonia event. Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Pneumonia will be scored according to the Utrecht Pneumonia Scoring System.

SECONDARY OUTCOMES:
Length of stay | Time between date of surgery and first discharge from ICU and first discharge from hospital (on average 14 days)
  Postoperative length of stay on the intensive care unit, Postoperative length of hospital stay.
Duration of mechanical ventilation | Time between intubation and first extubation (in general no more then 24 hours)
  Number of hours spent on the mechanical ventilator during and directly following the primary surgery.
Respiratory muscle function | At baseline, before surgery and 3, 6 and 9 days after surgery.
  Inspiratory muscle endurance and maximal inspiratory pressure at the mouth (Pi-max).
Pulmonary function | At baseline, before surgery and 3, 6 and 9 days after surgery.
  Forced Expiratory Volume in one second (FEV1), Forced vital capacity (FVC), FEV1/FVC ratio.
Quality of life | At baseline and 4 weeks after surgery
  Quality of life is measured using the EuroQol and SF-12 questionnaires.

CONTACTS AND LOCATIONS:
Locations (9):
- University Hospital Gasthuisberg, Leuven, Belgium
- HUS, Helsinki, Finland
- St. James's Hospital, Dublin, Ireland
- Netherlands (6):
  - Zorggroep Twente, Almelo
  - VU Medical Center, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Atrium Medical Center, Heerlen
  - Canisius Wilhelmina Hospital, Nijmegen
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Valkenet K, Trappenburg JCA, Ruurda JP, Guinan EM, Reynolds JV, Nafteux P, Fontaine M, Rodrigo HE, van der Peet DL, Hania SW, Sosef MN, Willms J, Rosman C, Pieters H, Scheepers JJG, Faber T, Kouwenhoven EA, Tinselboer M, Rasanen J, Ryynanen H, Gosselink R, van Hillegersberg R, Backx FJG. Multicentre randomized clinical trial of inspiratory muscle training versus usual care before surgery for oesophageal cancer. Br J Surg. 2018 Apr;105(5):502-511. doi: 10.1002/bjs.10803. PMID 29603130
- [Derived] Valkenet K, Trappenburg JC, Gosselink R, Sosef MN, Willms J, Rosman C, Pieters H, Scheepers JJ, de Heus SC, Reynolds JV, Guinan E, Ruurda JP, Rodrigo EH, Nafteux P, Fontaine M, Kouwenhoven EA, Kerkemeyer M, van der Peet DL, Hania SW, van Hillegersberg R, Backx FJ. Preoperative inspiratory muscle training to prevent postoperative pulmonary complications in patients undergoing esophageal resection (PREPARE study): study protocol for a randomized controlled trial. Trials. 2014 Apr 27;15:144. doi: 10.1186/1745-6215-15-144. PMID 24767575